CLINICAL TRIAL: NCT04275102
Title: A Feasibility Study of Three Times Weekly Symptom Screening for Children With Cancer
Brief Title: Three Times Weekly Symptom Screening for Children With Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Lillian Sung, Principal Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REB# 1000063548
Record Dates: First submitted 2019-12-11; First posted 2020-02-19 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Relapsed Cancer
MeSH Terms: conditions — Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Three times weekly symptom screening (Experimental): Three times weekly symptom reporting by guardians and children using the SPARK platform for 8 weeks
  Interventions: Other: SPARK

INTERVENTIONS:
Other: SPARK — Prompt to complete symptom screening three times weekly via SPARK with corresponding feedback sent to healthcare providers with each completed assessment.

SUMMARY:
This study will evaluate the feasibility of three times weekly symptom reporting by children using the SPARK platform for 8 weeks. SPARK is a web-based application that promotes symptom screening for children receiving cancer therapies and enables access to clinical practice guidelines for symptom management. Newly diagnosed and relapsed patients with cancer will be enrolled. Children and/or their guardian will be prompted to complete symptom screening three times weekly via SPARK with corresponding feedback sent to their healthcare providers with each completed assessment. Symptom reports will contain links to clinical practice guidelines for symptom management. Active intervention will last for 8 weeks starting from the date of enrollment.

DETAILED DESCRIPTION:
Primary objective is to determine the feasibility of three times weekly symptom reporting by guardians and children using the SPARK platform for 8 weeks. Feasibility will be evaluated by compliance with symptom screening and the investigators anticipate that at least 75% can achieve compliance with at least 60% of symptom evaluations.

Newly diagnosed and relapsed patients with cancer 2-18 years of age will be enrolled Children will be prompted to complete symptom screening three times weekly via SPARK with corresponding feedback sent to their healthcare providers with each completed assessment. Symptom reports will contain links to clinical practice guidelines for symptom management. Active intervention will last for 8 weeks starting from the date of enrollment.

Patient-reported outcomes will be obtained at baseline, and weeks 4, and 8. These outcomes will include the Symptom Screening in Pediatrics Tool (SSPedi), Fatigue will be measured using PROMIS, and the Pediatric Quality of Life Inventory (PedsQL) 3.0 Acute Cancer Module. Data from health records will be abstracted for all enrolled participants to evaluate symptom documentation and intervention provision at times symptom screening is completed as well as emergency room visits, clinic visits and hospitalizations.

Analyses are descriptive. The investigators' primary outcome is feasibility, sample size justification will focus on having sufficient number of guardians and children to optimize study processes and to describe the number of completed symptom assessments. The investigators will enroll up to 20-30 children per site per cohort; it is anticipated the investigators can enroll this number over one year. The 95% confidence intervals assuming 60% compliance will be 36-81% and 41-77% for 20 and 30 participants respectively; this precision is adequate for research purposes. If it is found that the processes are not feasible, the data will be reviewed after the initial cohort and enact refined procedures to rectify the identified problems. In this case enrollment of another 20-30 children per site per cohort with the updated procedures for a total sample size of 40-60 participants per site.

Primary objective of feasibility of responsive respondent type will be to evaluate the feasibility of eliciting bothersome symptoms using co-SSPedi, mini-SSPedi, co-mini-SSPedi, SSPedi or proxy-SSPedi. We will include children with cancer who: (1) are 2-18 years of age at enrollment; (2) are English, French or Spanish speaking (SSPedi is validated in these languages); (3) have any cancer diagnosis regardless of relapse status (4) have received or have a plan to receive any chemotherapy, radiotherapy or surgery. Exclusion criteria will be cognitive disability or visual impairment (cannot see SPARK even with corrective lens).

The same procedures as above will be followed with the exception that 1) PRO outcomes will be PROMIS Fatigue, PROMIS Pain Interference, the Pediatric Nausea Assessment Tool and SSPedi; 2) A qualitative feedback interview will be administered at week 4 and week 8. 3) At each reminder to complete symptom screening, the participant can choose which type of SSPedi they wish to complete. We will track type of SSPedi used. Participants may be contacted in person, by email, text, or over the phone to ensure there are no technical barriers to completing SSPedi.

All statistics are descriptive. As our primary outcome is feasibility, sample size justification will focus on having sufficient number of children to optimize study processes and to describe the number of completed symptom assessments. We will enroll 20-30 children per site per cohort and anticipate we can enroll this number over one year. The 95% confidence intervals assuming 60% compliance will be 36-81% and 41-77% for 20 and 30 participants respectively; this precision is adequate for our purposes. If we find that our processes are not feasible we will review the data after the initial cohort and enact refined procedures to rectify the identified problems. In this case we will enroll another 20-30 children per site per cohort with the updated procedures for a total sample size of 40-60 participants per site.

The sample size calculation for the responsive respondent component will be the same as for the SSPedi feasibility study .

ELIGIBILITY:
Inclusion Criteria:

* cancer diagnosis
* 2-18 years of age at enrollment
* Child has received or a plan for any chemotherapy, radiotherapy or surgery
* Understands English, French or Spanish

Exclusion Criteria:

* Cognitive disability
* Visual impairment (cannot see SPARK even with corrective lens)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-11-29 (Estimated); Study Completion 2025-11-29 (Estimated)

PRIMARY OUTCOMES:
Feasibility of three times weekly symptom reporting by children using the SPARK platform for 8 weeks. | 8 weeks
  The primary endpoint is feasibility, defined as at least 75% achieving compliance with at least 60% of symptom evaluations among guardian and self-report populations.

SECONDARY OUTCOMES:
Symptom burden as measured by the total SSPedi score Total SSPedi symptom scores | Baseline and weeks 4, and 8
  Total SSPedi symptom which is the sum of each of the 15 SSPedi item's Likert scores, resulting in a total score that ranges from 0 (no bothersome symptoms) to 60 (worst bothersome symptoms). The recall period is yesterday or today (SSPedi).
QoL will be measured using the PedsQL 3.0 Acute Cancer Module | Baseline and weeks 4, and 8
  Quality of life will be measured using the Pediatric Quality of Life Inventory (PedsQL) 3.0 Acute Cancer Module. The minimum value on the scale is 0 and maximum value is 100. PedsQL uses reverse scoring thus a higher score indicates a better outcome.
Symptom documentation | Baseline and weeks 4, and 8
  Symptom documentation and intervention provision at each time point in which symptom assessment is performed will be abstracted from the health record.
Number of Patients' Emergency Department Visits, Unplanned Clinic Visits and Hospitalizations over the 8-week intervention | Baseline and weeks 4, and 8
  The number of emergency department visits and unplanned clinic visits and hospitalizations over the 8-week intervention period will be abstracted from the health record.
Fatigue | Baseline and weeks 4, and 8
  Fatigue will be measured using PROMIS. The recall period is the last 7 days. It is reliable and valid in children 5-18 years of age with cancer
Nausea as measured by the Pediatric Nausea Assessment Tool | Baseline and weeks 4, and 8
  The recall period is today and yesterday. It is valid in children 4 to 18.
Pain as measured by PROMIS Pain Interference | Baseline and weeks 4, and 8
  The recall period is the last 7 days. It is reliable and valid in children 5-18 years of age with cancer

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Sung, MD, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT04275102/Prot_000.pdf